CLINICAL TRIAL: NCT07198763
Title: Comparison Between Conventional Rehabilitation and Conventional Rehabilitation Through Dance in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Comparison Between Conventional Rehabilitation and Conventional Rehabilitation Through Dance in Patients With COPD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Rio de Janeiro State Research Supporting Foundation (FAPERJ) (Other Government); Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 255.321
Record Dates: First submitted 2025-09-12; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Pulmonary Disease (COPD), Chronic Obstructive; Dance Therapy; Dance
Keywords: Dance; Chronic Obstructive Pulmonary Disease; Muscle Strength; Quality of live; Rehabilitation
MeSH Terms: conditions — Lung Diseases; Pulmonary Disease, Chronic Obstructive | interventions — Dance Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups: one group will perform conventional pulmonary rehabilitation twice a week and the other group will perform conventional pulmonary rehabilitation once a week and dance rehabilitation on another day of the same week for a total duration 12 weeks.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rehabilitation Program (RP): Group 1 (Active Comparator): Pulmonary rehabilitation program for 2 days per week, lasting approximately 50 minutes, for 8 weeks.
  Interventions: Other: Conventional pulmonary rehabilitation
- Pulmonary rehabilitation through dance: Group 2 (Experimental): Pulmonary rehabilitation program through dance for 2 days per week, lasting approximately 50 minutes, for 8 weeks.
  Interventions: Other: Conventional pulmonary rehabilitation

INTERVENTIONS:
Other: Conventional pulmonary rehabilitation — After completing the assessments, participants will be randomly divided into two groups: Group 1, which will perform PR exercises and the Group 2, which will perform PR through dance. Both groups will have the interventions of pulmonary rehabilitation during approximately 50 minutes, for 8 weeks. The group 1 will perform five different exercises with resistance bands, with 3 sets of 1 minute each. Exercises will always begin with the lightest resistance band, and if more than 30 repetitions are observed in 1 minute, the resistance band will be replaced with one of the next highest resistance. The Group 2 will perform rehabilitation through dance using 2 different playlists. The music will be from nationally and internationally known artists. The steps will be based on the exercises performed in group 1 and will be incremented throughout each song and playlist. At the end of 8 weeks of intervention, the evaluative tests will be applied again.
  Other Names: Pulmonary rehabilitation; Dance; Dance therapy

SUMMARY:
Introduction: Chronic obstructive pulmonary disease (COPD) is recognized as one of the most relevant conditions worldwide, due to its high morbidity and mortality. Patients classified by GOLD as groups B and E are strongly encouraged to participate in pulmonary rehabilitation (PR) programs. Dance has been shown to be equally or, at times, more effective as a rehabilitation strategy when compared to other types of physical activity. Objective: To compare the effect of conventional rehabilitation and the effect of conventional rehabilitation added to dance in patients with COPD. Methods: This is a conventional randomized controlled clinical trial to be carried at the Piquet Carneiro University Polyclinic, Rio de Janeiro. Patients diagnosed with COPD will be evaluated. Eligible participants will complete specific questionnaires and tests. Finally, participants will be randomly divided into two groups: one group will perform conventional PR twice a week and the other group will perform rehabilitation through dance twice a week using 2 different playlists. The music will be from nationally and internationally known artists during 8 weeks. The evaluation tests will be repeated at the end of the intervention. Expected results: It is expected that the group of individuals with COPD who perform rehabilitation through dance will obtain greater and better results in relation to exercise capacity, QoL and peripheral muscle strength when compared to the group that will carry out the intervention consisting of two days of conventional PR.

Keywords: Dance; Chronic obstructive pulmonary disease; Muscle strength; Quality of life; Rehabilitation.

DETAILED DESCRIPTION:
Introduction: Chronic obstructive pulmonary disease (COPD) is recognized as one of the most relevant conditions worldwide, due to its high morbidity and mortality. Patients classified by GOLD as groups B and E are strongly encouraged to participate in pulmonary rehabilitation (PR) programs. Dance has been shown to be equally or, at times, more effective as a rehabilitation strategy when compared to other types of physical activity. Objective: To compare the effect of conventional rehabilitation and the effect of conventional rehabilitation added to dance in patients with COPD. Methods: This is a conventional randomized controlled clinical trial to be carried at the Piquet Carneiro University Polyclinic, Rio de Janeiro. Patients diagnosed with COPD, of both sexes, will be evaluated. Eligible participants will complete quality of life questionnaires - 36-item Short Form (SF-36), the COPD Assessment Test (CAT) and the Hospital Anxiety and Depression Scale (HADS).

Additionally, patients will undergo pulmonary function tests, including spirometry, in addition to the six-minute walk test (6MWT), the handgrip test and the one repetition maximum test (1RM test). Finally, participants will be randomly divided into two groups: one group will perform conventional PR twice a week and the other group will perform rehabilitation through dance twice a week using 2 different playlists. The music will be from nationally and internationally known artists during 8 weeks. The evaluation tests will be repeated at the end of the intervention. Expected results: It is expected that the group of individuals with COPD who perform rehabilitation through dance will obtain greater and better results in relation to exercise capacity, QoL and peripheral muscle strength when compared to the group that will carry out the intervention consisting of two days of conventional PR.

Keywords: Dance; Chronic obstructive pulmonary disease; Muscle strength; Quality of life; Rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for COPD;
2. Age group over 40 years old;
3. Both genders;
4. Absence of acute exacerbation in the last 30 days;
5. Patients who are regularly using their medications.

Exclusion Criteria:

1. Presence of comorbidities and cardiovascular, neurological, renal, metabolic or musculoskeletal disorders that prevent the performance of functional tests;
2. Advanced cancer;
3. Previous lung surgery;
4. Inability to understand functional tests or questionnaires applied;
5. Patients who, during the research, present an acute exacerbation of COPD, due to the time required for recovery;
6. Patients with results observed in the 6MWT <300m.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2025-09-07 (Actual); Primary Completion 2025-09-07 (Actual); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
Exercise capacity. | 8 weeks.
  Assessment of participants' exercise capacity using the 6MWT, before and after rehabilitation.

SECONDARY OUTCOMES:
Quality of life assessment. | 8 weeks.
  A quality of life assessment will be performed correlating both groups of participants of the COPD research. For this purpose, the Brazilian version of the quality questionnaire - the 36-item Short Form (SF-36) - will be used.
  The SF-36 is a multidimensional questionnaire with a total of 36 items. It covers eight domains: functional capacity, physical functioning, pain, general health, vitality, social functioning, emotional functioning, and mental health. Scores can range from 0 to 100. Higher scores indicate greater overall patient well-being.
Peripheral muscle strength. | 8 weeks.
  A peripheral muscle strength will be performed correlating both groups of participants of the COPD research. For this purpose, the 1 repetition maximum (1RM) test and handgrip strength will be used.
  To analyze the intensity of anaerobic exercise, the 1RM quadriceps muscle extension test using a load cell will be used.
  For the handgrip test, participants will be instructed to sit and use their dominant hand. They will then rest their dominant elbow on a table, maintaining a 90° angle, and squeeze the dynamometer as tightly as possible. The test will be performed three times, lasting approximately 3 to 5 seconds, and all participants will receive verbal encouragement throughout. The highest handgrip value will be used.
Depression and anxiety. | 8 weeks.
  A depression and anxiety assessment will be performed correlating both groups of participants of the COPD research. For this purpose, the Anxiety and Depression Scale - Hospital Anxiety and Depression Scale (HADS) will be used.
  The HADS is a scale that assesses an individual's likelihood of experiencing anxiety, depression, or both. It consists of 14 items, each with four response options and a possible score of 0, 1, 2, or 3. There are three categories for anxiety and depression: unlikely (0-7 points), questionable or doubtful (8-11 points), and probable (12-21 points). A higher score indicates a greater likelihood of experiencing either disorder. It is important to note that the HADS has a reliability of 0.68 for anxiety and 0.77 for depression and has been validated for Brazilian Portuguese.

CONTACTS AND LOCATIONS:
Overall Officials: Thaís F de Andrade Lima, L.X., Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
The data obtained in the evaluation form, as well as the tests and questionnaires carried out, may be shared.

REFERENCES:
- [Background] Kaya M, Gurses HN, Ucgun H, Okyaltirik F. Effects of creative dance on functional capacity, pulmonary function, balance, and cognition in COPD patients: A randomized controlled trial. Heart Lung. 2023 Mar-Apr;58:13-20. doi: 10.1016/j.hrtlng.2022.10.017. Epub 2022 Nov 3. PMID 36335909